CLINICAL TRIAL: NCT02262650
Title: Relative Bioavailability of Telmisartan and SR26334, the Main Metabolite of Clopidogrel, After Co-administration Compared to the Bioavailability of Telmisartan and SR26334 After p.o. Administration of 80 mg Telmisartan and 75 mg Clopidogrel Alone. A Four-way, Single Dose, Open, Randomised Crossover Study in 24 Healthy Male and Female Subjects
Brief Title: Relative Bioavailability of Telmisartan and SR26334 After Co-administration Compared to the Bioavailability of Telmisartan and SR26334 After Administration of Telmisartan and Clopidogrel Alone in Healthy Male and Female Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 502.457
Record Dates: First submitted 2014-10-10; First posted 2014-10-13 (Estimated); Last update posted 2014-10-13 (Estimated); Status verified 2014-10

CONDITIONS: Healthy
MeSH Terms: interventions — Telmisartan; Clopidogrel

ARMS (4):
- Telmisartan alone (Active Comparator)
  Interventions: Drug: Telmisartan
- Telmisartan + Clopidogrel (concomitantly) (Experimental)
  Interventions: Drug: Telmisartan; Drug: Clopidogrel
- Telmisartan + Clopidogrel (consecutively) (Experimental)
  Interventions: Drug: Telmisartan; Drug: Clopidogrel
- Clopidogrel alone (Active Comparator)
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Telmisartan
  Arms: Telmisartan + Clopidogrel (concomitantly); Telmisartan + Clopidogrel (consecutively); Telmisartan alone
Drug: Clopidogrel
  Arms: Clopidogrel alone; Telmisartan + Clopidogrel (concomitantly); Telmisartan + Clopidogrel (consecutively)

SUMMARY:
Study to investigate the relative bioavailability of concomitant administration of clopidogrel and telmisartan (Test 1) relative to the bioavailability of SR26334 alone (Reference 1), and relative to the bioavailability of telmisartan alone (Reference 2). And to investigate the bioavailability of SR26334 following administration of clopidogrel 30 minutes after intake of telmisartan (Test 2) relative to the bioavailability of SR26334 alone (Reference 1), and relative to the bioavailability of telmisartan alone (Reference 2)

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects according to the following criteria: based upon a complete medical history, the physical examination, vital signs (BP, HR), 12-lead ECG, clinical laboratory tests
* Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice (GCP) and local legislation
* Age >= 40 years
* Body Mass Index (BMI) >=18.5 and <=29.9 kg/m2
* Good venous status of forearms

Exclusion Criteria:

* Any finding of the medical examination (including blood pressure, heart rate, and electrocardiogram) deviating from normal and of clinical relevance
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunologic or hormonal disorders
* Surgery of gastrointestinal tract (except appendectomy)
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of relevant orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of an allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* Intake of drugs with a long half-life (> 24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial
* Use of any drugs, which might reasonably influence the results of the trial based on the knowledge at the time of protocol preparation within 10 days prior to administration or during the trial
* Participation in another trial with an investigational drug within two months prior to administration or during the trial
* Smoker (more than 10 cigarettes or three cigars or three pipes/day)
* Alcohol abuse (more than 60 g/day)
* Drug abuse
* Blood donation or loss of more than 400 mL within four weeks prior to administration or during the trial.
* Excessive physical activities (within five days prior to administration or during the trial)
* Any laboratory value outside the reference range of clinical relevance
* History of hereditary fructose intolerance
* Veins unsuited for i.v. puncture on either arm (e.g. veins which are difficult to locate, access or puncture, veins with a tendency to rupture during or after puncture, etc.)
* Inability to comply with the dietary regimen of study centre
* Inability to comply with the investigators instructions

For female subjects:

* Pregnancy
* Positive pregnancy test
* No adequate contraception e.g. oral contraceptives, sterilization, intrauterine device (IUD)
* Inability to maintain this adequate contraception during the whole study period
* Lactation period

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2004-04; Primary Completion 2004-05 (Actual)

PRIMARY OUTCOMES:
AUC0-∞ (area under the concentration time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | up to 72 hours post dose
Cmax (maximum concentration of the analyte in plasma) | up to 72 hours post dose

SECONDARY OUTCOMES:
Number of subjects with adverse events | up to 8 days after last drug administration
Number of subjects with clinically significant findings in vital signs | up to 8 days after last drug administration
Number of subjects with clinically significant findings in ECG | up to 8 days after last drug administration
Number of subjects with clinically significant findings in labortory test | up to 8 days after last drug administration
tmax (time from dosing to the maximum concentration of the analyte in plasma) | up to 72 hours post dose
AUC0-tz (area under the concentration-time curve of the analytes in plasma over the time interval from 0 to the time of the last quantifiable data point) | up to 72 hours post dose
λz (terminal rate constant in plasma) | up to 72 hours post dose
t1/2 (terminal half-life of the analytes in plasma) | up to 72 hours post dose
MRTpo (mean residence time of the analytes in the body after po administration) | up to 72 hours post dose
CL/F (apparent clearance of the analytes in the plasma after extravascular administration) | up to 72 hours post dose
Vz/F (apparent volume of distribution during the terminal phase λz following an extravascular dose) | up to 72 hours post dose
CLR, 0-24 (renal clearance of SR26334 in plasma from the time point t1 until the time point t2) | up to 72 hours post dose